CLINICAL TRIAL: NCT01698125
Title: Autonomic Cardiovascular Control for Elderly Surgery Patients
Status: Terminated | Type: Observational
Why Stopped: Practical circumstances made it too difficult to carry out as planned.
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/2498/REK nord
Record Dates: First submitted 2012-09-27; First posted 2012-10-02 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Delirium
Keywords: Delirium; Autonomic cardiovascular control; Abdominal surgery; Tilt-test
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum. Plasma. Saliva.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abdominal surgery: Patients 65 years or older scheduled for abdominal surgery at Oslo University Hospital
  Interventions: Procedure: Abdominal surgery

INTERVENTIONS:
Procedure: Abdominal surgery — Patients 65 years or older scheduled for abdominal surgery at Oslo University Hospital

SUMMARY:
The purpose of this study is to study aspects of autonomic cardiovascular control and the level of stress hormones and inflammatory markers in saliva or serum, in elderly patients exposed to elective, major abdominal surgery, with or without postoperative delirium, to explore the hypothesis that delirium may be the result of aberrant stress responses.

DETAILED DESCRIPTION:
Patients admitted for elective, major, abdominal surgery will be tested with a head-up tilting to 20 degrees for 15 minutes preoperatively and again on the second postoperative day. Haemodynamic variables will be registered by the device TaskForceMonitor which monitors heart rate (HR), electrocardiography (ECG), blood pressure and stroke volume continuously and non-invasively.

Background variables (including demographics, comorbidity and simple cognitive tests) and daily variables (including delirium assessments) will be registered.

Blood and saliva samples will be drawn preoperatively and postoperatively to measure levels of stress hormones and inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years or older scheduled for abdominal surgery at Oslo University Hospital

Exclusion Criteria:

* Absence of a valid informed consent or assent, or consent from a legal proxy
* Patients with atrial fibrillation or a pacemaker rhythm
* Polyneuropathy
* Current treatment with beta-blockers, calcium-blockers or cholinesterase inhibitors
* Competing research project

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients scheduled for abdominal surgery at Oslo University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in orthostatic cardiovascular responses | Baseline and postoperatively at surgical ward (expected second postoperative day)
  Change in orthostatic cardiovascular responses (head-up tilt test) pre- and postoperatively in patients with and without postoperative delirium will be evaluated based on measurements of heart rate, systolic blood pressure (BP), mean BP, diastolic BP, stroke index, total peripheral resistance index, end-diastolic volume index, and acceleration index.

SECONDARY OUTCOMES:
Barthel Activities of Daily Living (ADL) Scale | Baseline
  Score from 0-20 points
Nottingham Extended Activity of Daily Living (NEADL) Scale | Baseline
  Score from 0-66 points.
Cumulative Illness Rating Scale | Baseline
  Total score from 0-56.
Dementia | Baseline
  Simple cognitive tests preformed preoperatively, including MMSE, Clock Drawing Test, Trail making A and B and Ten word memory test. Also IQCODE when reliable information is present.
Delirium | Baseline and a minimum of 2 days after the second tilt-test, an expected average of 5 days.
  Daily assessing the patient using the Confusion Assessment Method (CAM), shortened version.
Cortisol | Baseline and second postoperative day
  Looking for differences in levels of cortisol in saliva (morning samples) pre-and postoperatively in patients developing delirium compared to patients not developing delirium.
Severity of delirium | Baseline and a minimum of 2 days after the second tilt-test, an expected average of 5 days
  Daily assessing the patient using MDAS (the memorial delirium assessment scale). Total score from 0-30.
Gait speed | Baseline
  Measuring comfortable gait speed at length of 4 meters, best result of 2 tests. Result in meter per second.

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir B Wyller, MD, Prof, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Ullevaal, Oslo, Norway